CLINICAL TRIAL: NCT06806371
Title: PREDICTORS of CARDIOVASCULAR OUTCOMES in INDIVIDUALS with DIFFERENT OBESITY PHENOTYPES
Acronym: PRE-CAR
Status: Active, not recruiting | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 401432
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this observational study is to identify and evaluate adverse cardiovascular outcomes in metabolically healthy obese individuals in a cohort of 25 to 64 years of age, both men and women. The main questions it aims to answer are: what are the markers of adverse cardiovascular outcomes in metabolically healthy obese individuals?

DETAILED DESCRIPTION:
The study is planned to include 1,600 people of the Ryazan city population aged 25-64 years, selected using a three-stage cluster sampling method. Participation in the study is voluntary, as evidenced by the signing of informed consent. Among them, it is planned to select obese people and conduct phenotyping according to the criteria of the National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III).

It is planned to conduct a survey at all stages of the study. The questionnaire will include the following modules: social status, dietary habits (dietary habits), physical activity, smoking, alcohol consumption, family history, personal history, objective data, laboratory data, data on medical care and disability, quality of life questionnaire. Measurement of blood pressure, heart rate, height, weight, waist circumference. Laboratory tests: total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides, glucose, fibrinogen, uric acid, C-reactive protein (by quantitative method).

Next, it is planned to monitor the examined individuals and collect endpoints for 36 months. The endpoints are: death from any cause, stroke of any etiology, fatal and non-fatal myocardial infarction and coronary artery revascularization, carotid artery surgery. Next, it is planned to establish a relationship between the studied indicators and the frequency of adverse outcomes in individuals with different obesity phenotypes.

ELIGIBILITY:
Inc1. Body mass index >=30 kg/m2 . 2. Less than three of the five criteria according to The National Cholesterol Education Program's Adult Treatment Panel III, NCEP/ATP III):

* Systolic blood pressure >130 and/or diastolic blood pressure >85 mmHg,
* Triglycerides >1.7 mmol/L,
* High density lipoproteins < 1.03 (men), < 1.29 (women);
* fasting plasma glucose >=5.6 mmol/L,
* waist circumference >102 cm (men), >88 cm (women)lusion Criteria:

Exclusion Criteria:

The presence of

* signs of chronic heart failure,
* coronary heart disease,
* infiltrative or hypertrophic obstructive cardiomyopathy or constrictive pericarditis,
* heart disease or valve disease, which can be expected to lead to surgery during the study,
* cancer.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: city of Ryazan
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2027-12-29 (Estimated); Study Completion 2028-01-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse cardiovascular outcomes | From inclusion in the study to three years
  The number of people with the following adverse outcomes will be recorded: death from any cause, nonfatal myocardial infarction, nonfatal stroke, coronary artery revascularization, carotid artery surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander N Vorobiev, Candidate of Medical Sciences, Study Director — Ryazan State Medical University
Locations (1):
- Ryazan State Medical University, Ryazan, Russia

IPD SHARING:
Plan to Share IPD: Undecided
the amount of information is determined